CLINICAL TRIAL: NCT04321057
Title: Cardial-MASS-Study: Influencing Factors on Reliability of Selfreported Weight and Height in Patients With Cardiovascular Disease
Brief Title: Cardial-MASS-Study: Influencing Factors on Reliability of Selfreported Weight and Height
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: Cardial-MASS
Record Dates: First submitted 2020-03-20; First posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Group questionnaire: Patient's height and weight are asked by questionnaire in this group. It includes patients at the cardiological department of Saarland University.
- Group male doctor: Patient's height and weight are asked by a male doctor in this group. It includes patients at the cardiological department of Saarland University.
- Group female doctor: Patient's height and weight are asked by a female doctor in this group. It includes patients at the cardiological department of Saarland University.
- Group male nurse: Patient's height and weight are asked by a male nurse in this group. It includes patients at the cardiological department of Saarland University.
- Group female nurse: Patient's height and weight are asked by a female nurse in this group. It includes patients at the cardiological department of Saarland University.
- Group family doctor: Patient's height and weight are asked by questionnaire in this group. This is the control group,including patients at a family doctor.

SUMMARY:
Height and weight are important informations in clinical life. Medication is dosed by them and weight, especially overweight, is a risk factor for cardiovascular diseases. Mostly you have to rely on the self-reported informations, because there is plenty of work and little time to weigh and measure every patient. But can the investigators really trust this informations? Former studies have shown, that most of self-reported heights and weights differ from the measured ones. This fact might lead to a wrong dosage of medicine or underestimated risk factors. So the Cardial-MASS-Study tries to detect influencing factors on the reliability of self-reported informations especially among patients, treated at the cardiological department at Saarland University.

DETAILED DESCRIPTION:
Weight and height of patients is often recorded in clinical practice, as well as in clinical research. They give important informations for medication dosages, e.g., anticoagulants or anesthesias. Furthermore, the body mass index (BMI), calculated by weight and height, is an easy instrument to estimate a patient's risk for cardiovascular diseases based on obesity.

In clinical practice, informations about height and weight do often rely on self-reported values instead of measured ones. This can be due to limited timely, but also instrumental resources, when scales or measuring tapes are not available. Unfortunately, these self-reported informations are often inaccurate. Age, education, weight, and sex seam to influence and distort them in different ways.

Former studies have shown, that a lot of patients overestimate their height [1-8] and underestimate their weight [1-6]. This might lead to a wrong classification in normal weight and overweight using BMI. Among elderly (>60 years) informations relying on measured values and on self-reported values seem to be even more divergent [10].

People with overweight are tending to underestimate their weight stronger than people with normal weight. The higher the weight, the more the self-reported information deviates from the actual weight [11,12]. Men's informations are more exact than women's, like Niedhammer et al. has shown in a study with 7350 participants [9]. Men with a BMI lower than 25 even overestimated their weight. Compared to younger ones, elderly men underestimated their weight more often, and elderly women's self-reported weight was more accurate [1,9].

Next to age and gender, socioeconomic variables do influence self-reported measures. The higher the education or working position the more accurate the information about height. Noteworthy, women in high working positions overestimate their height, when compared to women in lower positions, who even underestimate their height [2,5,6,8,9].

Furthermore, external conditions of data acquisition may impact validity of self-reported information, too. Stewart supposed that informations given in an interview are more exact than those given in a questionnaire [11].

Most of the studies mentioned above are not exclusively related to patients with cardiovascular diseases. Studies referring to this patient population suggest, that men with cardiovascular diseases underestimate their weight less than others [13]. Nevertheless, Niedhammer et al. could not confirm this finding [9]. HEnce, the aim of this study is to identify factors that influence the validity of self-reported height and weight in patients with cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Innere Medizin III (Cardiology), Universitätsklinikum des Saarlandes (UKS)
* cardiovascular disease (Coronar-Vessel-Disease, Arrhythmia, Heart-attack, Hypertonus, stable heart failure)
* Patients at a family doctor

Exclusion Criteria:

* younger than 18 years
* Dementia
* cardial decompensation
* severe anemia (Hemoglobin<9 mg/dl)
* cardial shock
* acute kidney failure
* factors, that prevent patients from answering the questionnaire
* factors, that prevent patients from being measured and weighted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Innere Medizin III, who participate voluntarily and who suffer at least from one cardiovascular disease
Sampling Method: Non-Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported weight | baseline
  Patient´s self-reported weight and the measured weight will be compared.
Self-reported height | baseline
  Patient´s self-reported height and the measured height will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Internal Medicine, Cardioloy, Angioloy, and Internal Intensive Care Medicine, Saarland University Hospital, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palta M, Prineas RJ, Berman R, Hannan P. Comparison of self-reported and measured height and weight. Am J Epidemiol. 1982 Feb;115(2):223-30. doi: 10.1093/oxfordjournals.aje.a113294. PMID 7058781
- [Background] Stewart AL. The reliability and validity of self-reported weight and height. J Chronic Dis. 1982;35(4):295-309. doi: 10.1016/0021-9681(82)90085-6. No abstract available. PMID 7061685
- [Background] Millar WJ. Distribution of body weight and height: comparison of estimates based on self-reported and observed measures. J Epidemiol Community Health. 1986 Dec;40(4):319-23. doi: 10.1136/jech.40.4.319. PMID 3655624
- [Background] Stewart AW, Jackson RT, Ford MA, Beaglehole R. Underestimation of relative weight by use of self-reported height and weight. Am J Epidemiol. 1987 Jan;125(1):122-6. doi: 10.1093/oxfordjournals.aje.a114494. PMID 3788941
- [Background] Rowland ML. Self-reported weight and height. Am J Clin Nutr. 1990 Dec;52(6):1125-33. doi: 10.1093/ajcn/52.6.1125. PMID 2239790
- [Background] Bowlin SJ, Morrill BD, Nafziger AN, Jenkins PL, Lewis C, Pearson TA. Validity of cardiovascular disease risk factors assessed by telephone survey: the Behavioral Risk Factor Survey. J Clin Epidemiol. 1993 Jun;46(6):561-71. doi: 10.1016/0895-4356(93)90129-o. PMID 8501483
- [Background] Ziebland S, Thorogood M, Fuller A, Muir J. Desire for the body normal: body image and discrepancies between self reported and measured height and weight in a British population. J Epidemiol Community Health. 1996 Feb;50(1):105-6. doi: 10.1136/jech.50.1.105. No abstract available. PMID 8762365
- [Background] Bostrom G, Diderichsen F. Socioeconomic differentials in misclassification of height, weight and body mass index based on questionnaire data. Int J Epidemiol. 1997 Aug;26(4):860-6. doi: 10.1093/ije/26.4.860. PMID 9279620
- [Background] Niedhammer I, Bugel I, Bonenfant S, Goldberg M, Leclerc A. Validity of self-reported weight and height in the French GAZEL cohort. Int J Obes Relat Metab Disord. 2000 Sep;24(9):1111-8. doi: 10.1038/sj.ijo.0801375. PMID 11033979
- [Background] Kuczmarski MF, Kuczmarski RJ, Najjar M. Effects of age on validity of self-reported height, weight, and body mass index: findings from the Third National Health and Nutrition Examination Survey, 1988-1994. J Am Diet Assoc. 2001 Jan;101(1):28-34; quiz 35-6. doi: 10.1016/S0002-8223(01)00008-6. PMID 11209581
- [Background] Jalkanen L, Tuomilehto J, Tanskanen A, Puska P. Accuracy of self-reported body weight compared to measured body weight. A population survey. Scand J Soc Med. 1987;15(3):191-8. doi: 10.1177/140349488701500311. PMID 3616534
- [Background] Roberts RJ. Can self-reported data accurately describe the prevalence of overweight? Public Health. 1995 Jul;109(4):275-84. doi: 10.1016/s0033-3506(95)80205-3. PMID 7667492
- [Background] Jeffery RW. Bias in reported body weight as a function of education, occupation, health and weight concern. Addict Behav. 1996 Mar-Apr;21(2):217-22. doi: 10.1016/0306-4603(95)00050-x. PMID 8730524
- [Background] Bray GA. Overweight is risking fate. Definition, classification, prevalence, and risks. Ann N Y Acad Sci. 1987;499:14-28. doi: 10.1111/j.1749-6632.1987.tb36194.x. PMID 3300479
- [Background] Pi-Sunyer FX. Medical hazards of obesity. Ann Intern Med. 1993 Oct 1;119(7 Pt 2):655-60. doi: 10.7326/0003-4819-119-7_part_2-199310011-00006. PMID 8363192
- [Background] Lavie CJ, Milani RV, Ventura HO. Obesity and cardiovascular disease: risk factor, paradox, and impact of weight loss. J Am Coll Cardiol. 2009 May 26;53(21):1925-32. doi: 10.1016/j.jacc.2008.12.068. PMID 19460605
- [Background] Kurth T, Gaziano JM, Berger K, Kase CS, Rexrode KM, Cook NR, Buring JE, Manson JE. Body mass index and the risk of stroke in men. Arch Intern Med. 2002 Dec 9-23;162(22):2557-62. doi: 10.1001/archinte.162.22.2557. PMID 12456227
- [Background] Dorn JM, Schisterman EF, Winkelstein W Jr, Trevisan M. Body mass index and mortality in a general population sample of men and women. The Buffalo Health Study. Am J Epidemiol. 1997 Dec 1;146(11):919-31. doi: 10.1093/oxfordjournals.aje.a009218. PMID 9400333
- [Background] Bender R, Trautner C, Spraul M, Berger M. Assessment of excess mortality in obesity. Am J Epidemiol. 1998 Jan 1;147(1):42-8. doi: 10.1093/oxfordjournals.aje.a009365. PMID 9440397
- [Background] Coe TR, Halkes M, Houghton K, Jefferson D. The accuracy of visual estimation of weight and height in pre-operative supine patients. Anaesthesia. 1999 Jun;54(6):582-6. doi: 10.1046/j.1365-2044.1999.00838.x. PMID 10403874
- [Background] Hendershot KM, Robinson L, Roland J, Vaziri K, Rizzo AG, Fakhry SM. Estimated height, weight, and body mass index: implications for research and patient safety. J Am Coll Surg. 2006 Dec;203(6):887-93. doi: 10.1016/j.jamcollsurg.2006.08.018. Epub 2006 Oct 25. PMID 17116557
- [Background] Foil MB, Collier MS, MacDonald KG Jr, Pories WJ. Availability and Adequacy of Diagnostic and Therapeutic Equipment for the Morbidly Obese Patient in an Acute Care Setting. Obes Surg. 1993 May;3(2):153-156. doi: 10.1381/096089293765559494. PMID 10757911
- [Derived] Therre M, Kindermann I, Wedegartner SM, Gross S, Schwantke I, Mahfoud F, Bohm M. Determinants of reliability of self-reported height and weight and their impact on medication dosing: a cross-sectional study. BMJ Open. 2025 Apr 15;15(4):e090020. doi: 10.1136/bmjopen-2024-090020. PMID 40233951